CLINICAL TRIAL: NCT06013254
Title: Effect of Sour Liquid On Swallowing Function of the Patients With Post-Stroke Dysphagia
Brief Title: Effect of Sour Liquid On Swallowing Function of the Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Ozgul Erol, Professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TÜTF-BAEK 2021/214
Record Dates: First submitted 2023-08-15; First posted 2023-08-28 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Acute Stroke
Keywords: acute stroke; dysphagia; swallowing function; sour taste
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 4 ml of freshly squeezed lemon juice with a pH of 2.8 at room temperature was administered under the supervision of the physician before breakfast, lunch, and dinner for patients with ischemic stroke. For patients with severe swallowing disorders according to the GUSS, lemon juice was administered using a syringe, drop by drop, at a volume of 4 ml over approximately 15-20 minutes, as tolerated by the patient, under the supervision of the physician. Patients with severe swallowing disorders were unable to swallow and consequently drooled the lemon juice out of their mouths. This procedure was continued for seven days.
  Interventions: Dietary Supplement: sour liquid
- Control group (No Intervention): 4 ml of room temperature water was administered under the supervision of the physician before breakfast, lunch, and dinner. For patients with severe swallowing disorders according to the GUSS, water was administered using a syringe, drop by drop, at a volume of 4 ml over approximately 15-20 minutes, as tolerated by the patient, under the supervision of the physician. Patients with severe swallowing disorders were unable to swallow and consequently drooled the water out of their mouths. This procedure was continued for seven days.

INTERVENTIONS:
Dietary Supplement: sour liquid — applying lemon juice
  Arms: Intervention group

SUMMARY:
The aim of this study was to evaluate the effect of early administration of sour liquid on swallowing function of patients with post-stroke dysphagia.

Hypothesis of the study were; H0: The sour liquid given early to patients with post-stroke dysphagia does not have an effect on swallowing function H1: The sour liquid given early to patients with post-stroke dysphagia has an effect on swallowing function The data of the study were collected using the "Personal Information Form," "Standard Swallowing Test," "Gagging Swallowing Screening Test (GUSS)," and the " National Institute of Health Stroke Scale (NIHSS)".

Early administration of sour liquid to patients with post-stroke dysphagia was found to have a positive effect on swallowing function.

DETAILED DESCRIPTION:
Background: Untreated and undetected swallowing disorders lead to increased morbidity and mortality in acute stroke patients due to inadequate nutrition, dehydration, and aspiration pneumonia leading to prolonged hospital stays, decreased functionality, and increased long-term care needs. The aim of this study was to evaluate the effect of early administration of sour liquid on swallowing function of patients with post-stroke dysphagia.

Materials and methods: This study was a randomized controlled trial, which was conducted with 95 patients with confirmed diagnosis of ischemic stroke and dysphagia, admitted to the neurology department of a university hospital. The intervention group (n=47) received 4 ml of room temperature lemon juice, while the control group (n=48) received 4 ml of room temperature water before breakfast, lunch, and dinner for a duration of 7 days. The Standard Swallowing Test, Gagging Swallowing Screen, and National Institutes of Health Stroke Scale were applied. Swallowing function and stroke severity were assessed at initial assessment, at the end of the 7th and 30th days.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with ischemic stroke,
* had not completed the first 72 hours after diagnosis,
* developed swallowing disorders,
* volunteered to participate in the study

Exclusion Criteria:

* diagnosed hemorrhagic stroke,
* had completed the first 72 hours after diagnosis,
* not developed swallowing disorders,
* not volunteered to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-11-20 (Actual)

PRIMARY OUTCOMES:
swallowing assessments using the Gugging Swallowing Screen (GUSS) score | initial assessment, 7th day assessment, 30th day assessment
  improve the swallowing disorders of patients who have experienced acute stroke through the administration of sour taste. patients in both the intervention and control groups underwent advanced swallowing assessments using the GUSS.
  Gugging Swallowing Screen (GUSS)consists of two parts including an indirect swallowing test with three subtests, and a direct swallowing test with four subtests. Evaluation is made on a scale of 0-20 as follows: 0-9 points indicate severe swallowing disorder with high risk of aspiration, 10-14 points indicate moderate swallowing disorder with moderate risk of aspiration, 15-19 points indicate mild swallowing disorder with low risk of aspiration, and 20 points indicate no swallowing disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Sezgin Kehaya, MD, Principal Investigator — Doctor of Neurology Clinic
Locations (1):
- Trakya University Faculty of Medicine, Edirne, Turkey (Türkiye)